CLINICAL TRIAL: NCT04706286
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety of CKD-393 and Co-administration of CKD-501, D759 and D150 Under Fed Condition in Healthy Adults
Brief Title: Clinical Trial to Investigate the Pharmacokinetics and Safety of CKD-393
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A98_03BE2018
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 1. Period 1: Treatment A
  2. Period 2: Treatment B
  Interventions: Drug: CKD-501, D759, D150; Drug: CKD-393 0.5/100/1000 mg
- Group 2 (Experimental): 1. Period 1: Treatment B
  2. Period 2: Treatment A
  Interventions: Drug: CKD-501, D759, D150; Drug: CKD-393 0.5/100/1000 mg

INTERVENTIONS:
Drug: CKD-501, D759, D150 — CKD-501 0.5 mg 1T, D759 100 mg 1T and D150 1000 mg 1T, single oral administration under fed condition
  Other Names: Treatment A
Drug: CKD-393 0.5/100/1000 mg — CKD-393 0.5/100/1000 mg 1T, single oral administration under fed condition
  Other Names: Treatment B

SUMMARY:
A Clinical Trial to evaluate the Pharmacokinetics and safety of CKD-393 0.5/100/1000 mg under fed condition

DETAILED DESCRIPTION:
A Phase 1 Clinical Trial to evaluate the safety and pharmacokinetics in healthy adult volunteers after administration of CKD-393 0.5/100/1000 mg under fed condition.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult who is 19 ~ 55 years at the time of screening
2. Body weight more than 55 kg for male and more than 50kg for female
3. BMI more than 18.5 kg/m2 or less than 27.0 kg/m2
4. Females must be menopause or surgical infertility
5. Males who have consented to the use of appropriate pregnancy contraceptive methods up to 28 days after the last investigational product and not to provide sperm
6. Subjects who voluntarily decided to participate and informed consent based upon understanding on the study.

Exclusion Criteria:

1. Subjects who have a history of clinically significant hepatic, renal, nervous, immune, respiratory, urinary, digestion, endocrine, hematooncology, cardiovascular systemic disease or psychosis disorder
2. Subjects who have genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
3. Subjects with poor oral intake, susceptible to dehydration or clinically significant dehydration
4. Subjects who have a history of gastrointestinal disorders (Crohn's disease, ulcerative colitis, etc.) or surgery (except simple appendectomy or hernia surgery) that may affect the absorption of the drug
5. Subjects who have a history of clinically significant hypersensitivity to drugs or additives
6. Subjects who have severe infectious disease and severe trauma before and after operation
7. Subjects who have undergone i.v. testing of radioactive iodine contrast material within 48 hours before the first IP administration
8. Subjects who are deemed unsuitable as subjects in the screening test performed within 28 days before the administration of investigational product

   * AST, ALT> UNL(Upper Normal Limit)x1.25
   * eGFR (Estimated Glomerular Filtration Rate) <60 mL/min/1.73m2 using the MDRD (Modification of Diet in Renal Disease) equation
   * Positive immunologic serological tests (hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test, syphilis test)
   * After resting for more than 5 minutes, systolic blood pressure> 150 mmHg or < 90 mmHg, diastolic blood pressure> 100 mmHg or <50 mmHg
9. Subjects who have had a history of drug abuse within one year of screening or have tested positive on urine drug screening test
10. Subjects who judged to able to affect in the study or in the subject's safety by the investigator for the following reasons

    * Ethical-the-counter (ETC) drugs and herbal medicines within 14 days of the first administration of the investigational drug.
    * Over-the-counter (OTC) drugs, including health foods and vitamin preparations, within 7 days of the first dose of the investigational product
    * Inducing or inhibiting drugs of drug-metabolism enzyme, within 30 days of the first dose of the investigational product
11. Subjects who have consistently excessively smoked or consumed caffeine or alcohol (caffeine:> 5 cups / day, alcohol:> 210 g / week, cigarettes:> 10 cigarettes / day) or cannot stop smoking, consuming caffeine and alcohol during hospitalization
12. Subjects who take grapefruit-containing food within 7 days before IP administration, or cannot forbid taking grapefruit-containing food for period of clinical trials.
13. Subjects who have received the investigational product by participating in other clinical trials (including bioequivalence studies) within 180 days before the first dose of the investigational product (For biological agents, this may be based on a longer period of time, considering the half-life)
14. Subjects who donated whole blood within 60 days before the first dose of the investigational product or donated component blood donation within 30 days
15. Subjects who received a blood transfusion within 30 days before the first dose of the investigational product
16. Pregnant or lactating women
17. Subjects who were deemed to be inappropriate to participate in the study by the investigator judgment

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-02-18 (Estimated); Primary Completion 2021-03-29 (Estimated); Study Completion 2021-04-05 (Estimated)

PRIMARY OUTCOMES:
AUCt(Area Under Curve last) of CKD-393 | From predose, upto 48 hours post-dose
  Area under the plasma concentration time curve of CKD-393, from time zero up to the last measurable concentration.
Cmax of CKD-393 | From predose, upto 48 hours post-dose
  The maximum concentration observed of CKD-393 over blood sampling time.

CONTACTS AND LOCATIONS:
Overall Officials: Choon Ok Kim, M.D., Ph.D., Principal Investigator — Severance hospital of the Yonsei University
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No